CLINICAL TRIAL: NCT06368570
Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During Routine Cesarean Delivery to Inform Anesthetic Practice. a Prospective Patient-centred Multidisciplinary Mixed-method (PAS-EDU-RCD)
Brief Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During Routine Cesarean Delivery
Acronym: PAS-EDU-RCD
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24-04
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Well-Being, Psychological
Keywords: cesarean delivery; patient experience; neuraxial anesthesia
MeSH Terms: conditions — Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cesarean delivery with neuraxial anesthesia.: Patients who have a scheduled cesarean delivery with neuraxial anesthesia.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed by the research team to learn about their experience of Cesarean delivery with neuraxial anesthetic
  Other Names: Interview questions

SUMMARY:
This study aims to explore the experience that the patient has as they undergo a routine Cesarean Delivery (CD). The indication for undergoing a routine CD varies amongst patients, but usually there is either an obstetric or medical reason for requiring a planned delivery of an infant via CD. Similarly, the experience of the CD varies significantly between patients as there are many patient, surgical and anesthetic factors that interact to create the unique experience each patient has. This study aims to explore the patients' perspective and learn about their preferences, concerns and suggestions regarding their experience of CD and to then use this information to enhance the quality of future anesthesia care for elective CD.

Patients who have undergone a routine CD will be approached the day following their delivery, while their recollection of their experience is still fresh, and given the opportunity to participate in the study, which will involve the completion of a questionnaire as well as an interview lasting approximately 20-25 minutes. In addition to interviewing the patients, the study will also involve several interviews of obstetricians, anesthesiologists and nurses with the goal of seeing how the patients' experiences compare to the providers' perspective of the care they are delivering. Following the gathering of this information and identification of potential improvements in current practice a follow up study will be performed aiming to implement changes and improve the quality of anesthesia care during elective CD.

DETAILED DESCRIPTION:
Elective CD is predominantly performed under neuraxial anesthesia that allows patients to be awake and able to experience childbirth along their support person. There is a high maternal satisfaction associated with being able to experience childbirth, however there is also high incidence of anxiety associated with being aware of the surgical procedure that is occurring while under neuraxial anesthesia. There are a limited number of studies that have explored the experience of the patient while undergoing elective CD under neuraxial anesthesia and even fewer that have focused on the patient's perspective, that is used to educate health care professionals on how to improve the quality of anesthesia care during elective CD. This study aims to embrace the patient perspective to guide quality improvement in the delivery of elective CD.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* ASA Physical Classification Score II or III
* elective CD (i.e. scheduled between 7am - 5pm) as per institutional standards (see below)
* patients who underwent the additional procedure of tubal ligation, salpingectomy or myomectomy (of uterine fibroid <4cm) at the time of CD will be included as these are considered minor additional procedures

Exclusion Criteria:

* under 18 years of age
* unable to answer questions due to a language barrier or their mental state
* BMI at the time of delivery that falls in the super-morbidly obese category (BMI > 55m-2)
* Patients who have underwent preterm delivery (under 37 weeks gestation), had a multiple gestation pregnancy or if there was presence of a significant fetal anomaly
* Anesthetic technique that significantly deviates from the institutional standards (see below*) including patients who underwent elective CD under epidural or dural puncture epidural (DPE) technique
* Performance of myomectomy with fibroid size >4cm at the time of CD
* Patients who underwent emergent CD as well as those who had contraindicated or failed neuraxial anesthesia and required general anesthesia for or during their CD will also be excluded.

  * Institutional standards: spinal or combined spinal and epidural (CSE) with the standard dose of 1.8mL heavy bupivacaine 0.75% combined with intrathecal morphine 100-150 micrograms and fentanyl 10-15 micrograms. Administration of crystalloid co-loading at 10-15mL/kg following establishment of neuraxial and vasopressors (phenylephrine, norepinephrine or ephedrine) to maintain systolic blood pressure at baseline. Routine administration of acetaminophen (PR), ketorolac (IV), dexamethasone and ondansetron, unless contraindicated.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who deliver by scheduled cesarean section with neuraxial anesthesia at Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Patient questionnaire | Following scheduled c-section delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be asked to rate their experience of having a cesarean delivery with neuraxial anesthesia, in terms of satisfaction and their experience with any discomfort.
  Some questions are yes/no, some are on a scale from 1-10, where 1 = not at all and 10 = totally agree, and some are open-ended.
  The questionnaire will take approximately 10 minutes to complete.
Patient interview | Following scheduled c-section delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be interviewed in person by a member of the research team and asked open ended questions. Interviews will be recorded, transcribed and coded for themes.
  Responses are not reported on any scale. The interview will take approximately 30 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Nabecker, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No